CLINICAL TRIAL: NCT04854681
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TQB2928 Injection in Patients With Advanced Solid Tumors or Hematological Malignancies
Brief Title: Phase 1 Trial of the TQB2928 Injection in Patients With Advanced Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2928-I-01
Record Dates: First submitted 2021-04-21; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Tumors and Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2928 injection (Experimental): Dose Escalation: intravenous (IV) infusion of TQB2928 as monotherapy
  Interventions: Drug: TQB2928 Injection

INTERVENTIONS:
Drug: TQB2928 Injection — 4 weekly IV infusions (Days 1, 8, 15, and 22) of TQB2928 in each 28-day treatment cycle until unacceptable toxicity, documentation of confirmed progressive disease (PD), or subject withdrawal.

SUMMARY:
TQB2928 is a promising new molecular entity that mediates blockade of CD47 and SIRPα and enhances the phagocytosis of cancer cells by macrophages. In preclinical in vivo models, TQB2928 was active against a wide range of solid tumors and hematologic malignancies. This is the first-in-human phase 1 trial of TQB2928 in patients with advanced solid tumors and hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.

  2. Histologically or cytologically confirmed, locally advanced unresectable or metastatic solid tumors, or hematological malignancies, or lymphoma.

  3. Solid tumors or hematological malignancies that failed from standard therapy, or lymphoma patients who have had at least two regimens of systemic therapy failures, or who refused other systemic therapy.

  4. At least 1 measurable lesion according to tumor-appropriate response criteria.

  5. Must have adequate organ and bone marrow function. 6. Resolved acute effects of any prior therapy to baseline severity or Grade ≤1 per CTCAE v5.0 except for AEs not constituting a safety risk by investigator judgment.

  7. Serum pregnancy test (for females of childbearing potential) negative within 7 days before enrollment.

  8. Male and female patients of childbearing potential and at risk for pregnancy must agree to use two highly effective method(s) of contraception throughout the study and for at least 90 days (180 days if required by local regulation) after the last dose of assigned treatment.

  9. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

* 1. Patients with known symptomatic brain metastases requiring steroids. 2. Concurrent secondary malignancy. 3. Uncontrolled pleural effusion or pericardial effusion with clinical significance and requiring repeated drainage as assessed by the Investigators.

  4. Prior treatment with monospecific or bispecific antibodies or fusion proteins targeting CD47 or signal regulatory protein alpha (SIRPα).

  5. Therapeutic or experimental monoclonal antibodies within 28 days prior to enrollment.

  6. Immunosuppressive regimens involving systemic corticosteroids (except <10 mg daily prednisone equivalent) within 14 days before the first dose of study treatment.

  7. Prior allogeneic hematopoietic stem cell transplant. 8. Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to enrollment.

  9. RBC transfusion dependence, defined as requiring more than 2 units of RBC transfusions during the 4-week period prior to screening. RBC transfusions are permitted during screening and prior to enrollment to meet the hemoglobin inclusion criteria.

  10. Vaccination within 4 weeks prior to enrollment except for administration of inactivated vaccines (for example, inactivated influenza vaccines) 11. Active and clinically significant bacterial, fungal or viral infection including tuberculosis, hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.

  12. History of hemolytic anemia or Evans syndrome within 3 months. 13. Autoimmune hemolytic anemia (AIHA) assessed by Positive Direct Antiglobulin Test (DAT).

  14. Autoimmune disorders (e.g., Crohn's Disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus) and other diseases that compromise or impair the immune system.

  15. Unstable or serious concurrent medical conditions in the previous 6 months. 16. Significant medical diseases or conditions, as assessed by the Investigators, that would substantially increase the risk-benefit ratio of participating in the study.

  17. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | During the first 28 days
  DLTs will be assessed during the first 28 days of treatment for dose-escalation and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (28 days) of treatment.
Maximum tolerated dose (MTD) | During the first 28 days
  MTD is defined as the highest dosing schedule cohort level at which no more than 1 of 6 patients experience a Dose Limiting Toxicity (DLT).

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) and serious adverse events (SAEs) | From the time of informed consent signed through 90 days after the last dose
  Assessed by CTCAE v5.0
Pharmacokinetics: Cmax | From the time of informed consent signed through 90 days after the last dose
  Maximum observed concentration (Cmax) of TQB2928 after administration
Pharmacokinetics: Cmin | From the time of informed consent signed through 90 days after the last dose
  Minimum observed concentration (Cmin) of TQB2928 at steady state
Pharmacokinetics: Tmax | From the time of informed consent signed through 90 days after the last dose
  Time to maximum concentration (Tmax)
Pharmacokinetics: AUC | From the time of informed consent signed through 90 days after the last dose
  The area under the curve (AUC) of serum concentration of TQB2928
Pharmacokinetics: T1/2 | From the time of informed consent signed through 90 days after the last dose
  Terminal half-life (T1/2)
Percentage of ADA positive patients | From the time of informed consent signed through 90 days after the last dose
  Number of patients who develop detectable anti-drug antibody (ADA), and percentage of ADA positive patients will be calculated to evaluate immunogenicity of TQB2928.
Objective Response Rate (ORR) | up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by iRECIST v1.1 criteria for solid tumors, Lugano2014 criteria and lymphoma response to immunomodulatory therapy criteria (LYRIC) for lymphoma, and AML IWG 2003 response criteria for acute myeloid leukemia (AML).
Disease control rate (DCR) | up to 2 years
  Defined as the proportion of subjects with CR, PR, or SD.
Duration of Response (DOR) | up to 2 years
  Defined as the time from first documented response to documented disease progression.
Progression-free survival (PFS) | up to 2 years
  Defined as the time from the first dose of TQB2928 to the first occurrence of disease progression or death from any cause.